CLINICAL TRIAL: NCT01984931
Title: Trimebutine Maleate (NEWBUTIN SR 300 mg Tab) as a Prophylactic Anti-emetic Drug for Patients Who Underwent Arthroscopic Rotator Cuff Repair: a Randomized Controlled Study
Brief Title: Study of Trimebutine Maleate (NEWBUTIN SR 300 mg Tab)for Treatment of Post Operative Nausea and Vomiting
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CM Chungmu Hospital (Other)
Collaborators: Korea United Pharm. Inc. (Industry)
Responsible Party: Principal Investigator, Sang-Hoon Lhee, Director of CM Chungmu Hospital, CM Chungmu Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CMH-2013-02
Record Dates: First submitted 2013-10-31; First posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Nausea; Vomiting
Keywords: post operative nausea and vomiting; Trimebutine Maleate
MeSH Terms: conditions — Nausea; Vomiting | interventions — Trimebutine; Bromazepam; mosapride; ruscogenin; Simethicone; lidaprim; Medazepam; Sunitinib; tricin; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trimebutine Maleate 300 mg Tab (Experimental): A single dose of NEWBUTIN SR 300 mg Tab will be given orally one hour prior to the said operation time and another 300 mg orally as soon as the patient wakes post operatively.
  Interventions: Drug: Trimebutine Maleate (NEWBUTIN SR 300 mg Tab)
- Metoclopramide hydrochloride monohydrate 8.46 mg/2ml/A (Active Comparator): Anti-emetic medication protocol of Chungmu Hospital includes MACPERAN (Metoclopramide hydrochloride monohydrate 8.46 mg/2ml/A)thru IV twice in a day
  Interventions: Drug: Metoclopramide hydrochloride monohydrate

INTERVENTIONS:
Drug: Trimebutine Maleate (NEWBUTIN SR 300 mg Tab) — Trimebutine Maleate (NEWBUTIN SR 300 mg Tab)is a noncompetitive spasmolytic agent. It possesses moderate opiate receptor affinity and has marked anti-serotonin activity especially on'M' receptors. A single dose of NEWBUTIN SR 300 mg Tab orally will be given one hour prior to the said operation time and another 300 mg orally as soon as the patient wakes post operatively.
  Other Names: •Antinime; •Cineprac; •Colixane B (Trimebutine and Bromazepam); •Colixane Prokin (Trimebutine and Mosapride); •Colixane; •Colonix B (Trimebutine and Bromazepam); •Colonix; •Colospasmyl; •Colperin; •Crobutin; •Debricol; •Debridat; •Débridat; •Eumotrix; •Ibuproct (Trimebutine and Ruscogenin); •Ibutin; •Libertrim; •Libertrim Pediátrico (pediatric); •Libertrim SDP (Trimebutine and Simeticone); •Libertrim SII (Trimebutine and Simeticone); •Muvett; •Polybutine; •Prescol; •Proctolog (Trimebutine and Ruscogenin); •Promebutin; •Ruscolog (Trimebutine and Ruscogenin); •Tribux; •Trimebutin; •Trimebutina Genfar; •Trimebutina La Santé; •Trimebutina; •Trimebutino Andromaco; •Trimedine; •Trimegam; •Trimet; •Altrip; •Apo-Trimebutine; •Biorgan B (Trimebutine and Bromazepam); •Biorgan; •Bumetin; •Butikinon; •Cerekinon; •Cerenamelin; •Colobutine; •Colypan; •Debretin; •Debricalm; •Debridat AP; •Debridat B (Trimebutine and Bromazepam); •Debridat Fort; •Debrum (Trimebutine and Medazepam); •Derispan; •Digerent; •Diway; •Dolpic; •Eumotil; •Eumotil-S (Trimebutine and Simeticone); •Eumotil-T (Trimebutine and Bromazepam); •Eutransil; •Fenatrop; •Garapepsin; •Gaspat; •Gismotal; •Liement; •Mebucolon; •Mebutit; •Miopropan; •Modulon; •Mustrick; •Muvett S (Trimebutine and Simeticone); •Newbutin SR; •Ni Wei Fu; •Pelkysil; •Pilemain; •Polibutin; •Recutin; •Rekelat; •Rui Jian; •Sakion; •Selumito; •Shuang Di; •Spabutine; •Spamoin; •Supeslone; •Sutent; •Tarabutine; •Tefmetin; •Tidomel; •Timotor; •Transacalm; •Tribudat Forte; •Tribudat; •Tributin; •Tricin; •Tridat; •Trienter; •Trim; •Trimebutin Maleate Taiyo; •Trimebutina Angenerico; •Trimebutina Colmed; •Trimebutina maleato; •Trimebutina MK; •Trimébutine Actavis; •Trimébutine Almus; •Trimébutine ALS; •Trimébutine Arrow; •Trimébutine Biogaran; •Trimébutine CristerS; •Trimébutine EG; •Trimébutine Evolugen; •Trimébutine Isomed; •Trimébutine maléate RPG; •Trimébutine Mylan; •Trimébutine Pfizer; •Trimébutine Qualimed; •Trimébutine Ranbaxy; •Trimébutine Ratio; •Trimébutine Ratiopharm; •Trimébutine Sandoz; •Trimébutine Teva; •Trimébutine Zentiva; •Trimébutine Zydus; •Trimebutino Maleato; •Trimedat; •Trishi; •VeM; •Yuan Sheng Li Wei
  Arms: Trimebutine Maleate 300 mg Tab
Drug: Metoclopramide hydrochloride monohydrate
  Arms: Metoclopramide hydrochloride monohydrate 8.46 mg/2ml/A

SUMMARY:
This study will determine if giving Trimebutine Maleate (NEWBUTIN SR 300 mg Tab)orally will be effective as a prophylactic anti-emetic drug for patients who underwent arthroscopic rotator cuff repair under general anesthesia.

DETAILED DESCRIPTION:
The patients will be divided in two groups using a computer generated randomization software. The first will be the MACPERAN group (controlled) and the other will be the NEWBUTIN group (variable). The controlled group will be treated with post-operative regimen in accordance with the standard protocol of the Chungmu Hospital, MACPERAN(Metoclopramide hydrochloride monohydrate 8.46 mg/2ml/A) thru IV twice in a day while the variable group will be given a single dose of NEWBUTIN SR 300 mg Tab orally one hour prior to the said operation time and another 300 mg orally as soon as the patient wakes post operatively.

A clinical research coordinator will monitor the patient until 48 hours post-operative. First time frame will be from 0-2 hours once patient is transferred to the ward followed by 2 hours to 24 hours and 24-48 hours post ward transfer. All patients will be assessed using the simplified risk score of Apfel et al. to determine who have the risk factors for PONV. The episodes of nausea and vomiting will be recorded taking note of its intensity and frequency on the said three time frames. Nausea is defined as a subjectively unpleasant sensation associated with an awareness of the urge to vomit; vomiting is defined as the forceful expulsion of gastric contents through the mouth. As retching is similar to vomiting in all aspects, except for the expulsion of gastric contents, it was considered as vomiting. The efficacy of anti-emetic medication (NEWBUTIN 300 mg/tab) will be assessed by monitoring the frequency and severity of nausea, vomiting, and PONV (which was regarded as the primary outcome). The severity of nausea will be graded on a four-point scale, where 0= no nausea, 1= mild nausea, 2= moderate nausea, and 3= severe nausea.Then the frequency will be assessed by monitoring how often the patient experienced these episodes (nausea and vomiting)during the said time frames.

ELIGIBILITY:
Inclusion Criteria:

* post arthroscopic cuff repair patient previously diagnosed with small to large rotator cuff tear thru MRI

Exclusion Criteria:

* above 70 years old
* massive rotator cuff tear

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-10; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Severity of nausea after taking Trimebutine Maleate as a prophylactic medication | 0-48 hours post rotator cuff repair
  The severity of nausea will be graded on a four-point scale. 0- no nausea (can do all tasks). 1- mild nausea (can talk and answer questions appropriately,sit, stand but can't walk). 2- moderate nausea (can talk and but answer questions inappropriately, sit but can't stand and walk). 3- severe nausea (don't talk and answer questions, prefers lying down, cannot sit, stand and walk).

SECONDARY OUTCOMES:
Frequency of PONV after taking Trimebutine Maleate as a prophylactic medication | 0-48 hours post rotator cuff repair
  Frequency is how often the patient experienced the episodes of nausea and vomiting in a given time period.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Alan B Tabar, MD, Principal Investigator — International Education Center of Shoulder, Elbow Surgery: Chungmu Hospital
Locations (1):
- Chungmu General Hopsital, Seoul, Yeongdeungpo-gu, South Korea